CLINICAL TRIAL: NCT00331123
Title: Study to Evaluate Efficacy and Safety of Transdermal Testosterone and Safety for an Open-label Period in Women With Hypoactive Sexual Desire Disorder on Estrogen Replacement Therapy and Undergone Hysterectomy/Bilateral Oophorectomy.
Brief Title: Study of Transdermal Testosterone Patches in Surgically Menopausal Women With Low Libido
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001133 and Yr 2-4 OL
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Surgical menopause; HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo
- Testosterone Patch (Experimental)
  Interventions: Drug: Testosterone Transdermal System

INTERVENTIONS:
Drug: Testosterone Transdermal System — testosterone patch, 300mcg/day, changed every 3-4 days for up to 52 weeks
  Arms: Testosterone Patch
Drug: Placebo — placebo patch,changed every 3-4 days for 24 weeks during double blind phase
  Arms: Placebo

SUMMARY:
This study is designed to evaluate efficacy and safety of a testosterone patch as treatment for low libido in surgically menopausal women who are taking estrogen therapy.

DETAILED DESCRIPTION:
Women with hypoactive sexual desire disorder (HSDD) who had undergone bilateral salpingo-oophorectomy and hysterectomy were randomized into a 52-week, multicenter, multinational study that included a 24-week, double-blind (DB), parallel-group, placebo-controlled period followed by a 28-week open-label (OL) period. Patients were stratified based on their use of oral or transdermal ET and randomized to receive placebo or testosterone transdermal system. Patients had to maintain a stable dose of estrogen throughout the study. Upon completion of the DB period, patients receiving placebo were switched to TTS, while the active cohort remained on active treatment. All patients were then followed for an additional 28 weeks for safety. Patients who completed the first 52 weeks of the study were given the opportunity to participate in an open label extension (Years 2, 3 , and 4), which was added to the protocol by amendment. Safety was assessed by adverse events, lipids, serum chemistry with hepatic, renal and carbohydrate metabolism evaluation, coagulation testing, and hematology. Physical exam including clinical assessments of facial hair and acne were monitored.

ELIGIBILITY:
Inclusion Criteria:

Eligible women must:

1. Be 20-70 years old and in generally good health
2. Have undergone hysterectomy and removal of both ovaries at least 6 months prior to screening
3. Be receiving a stable dose of estrogen replacement therapy for at least 3 months prior to screening with the intention of maintaining that regimen.
4. Be, in her own judgment, in a stable monogamous sexual relationship that is perceived to be secure and communicative, for at least one year prior to study entry.
5. Meet the criteria for having hypoactive sexual desire disorder.

Exclusion Criteria:

Eligible women must not:

1. Have received androgen therapy at any time during the past 3 months (during the past 7 months if therapy was an investigational implantable product)
2. Be experiencing any chronic or acute life stress relating to any major life change
3. Be experiencing depression and/or receiving medication for such illness or disorder
4. Have current severe skin problems (such as severe or cystic acne) or allergy to adhesives (like the ones in bandages)
5. Have had a major illness, active gall bladder disease, or gynecological or breast surgery within the last 6 months
6. Have a history of breast, endometrial, or other gynecological cancer any time before study participation or other cancer within the last 5 years
7. Have diabetes, a history of cerebrovascular disease, thromboembolic disorders, heart attack, or angina at any time before study participation or thrombophlebitis within the last 5 years
8. Have abnormal laboratory test results upon initial screening for this study
9. Have previously participated in P&GP study 1999068 or 1999092
10. Have previously participated in a clinical trial within 30 days or received an investigation medication within 30 days.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2002-05; Primary Completion 2003-12 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of testosterone transdermal system (TTS) as measured by the change from baseline in the frequency of total satisfying sexual activity captured by the Sexual Activity Log (SAL). | 24 weeks

SECONDARY OUTCOMES:
To assess the efficacy measured by the change from baseline in sexual desire; personal distress as measured by the Personal Distress Scale score; the other 6 domains of the profile of Female Sexual Function; and the other 8 SAL endpoints. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johna Lucus, MD, Study Director — Procter and Gamble
Locations (3):
- Research Site, Kansas City, Missouri, United States
- Research Site, Prahran, Victoria, Australia
- Research Site, Québec, Quebec, Canada